CLINICAL TRIAL: NCT07013396
Title: A Prospective Evaluation of Clinical Outcomes in Acute Ischemic Stroke After Endovascular Treatment Using Transcranial
Brief Title: A Prospective Evaluation of Clinical Outcomes in Acute Ischemic Stroke After Endovascular Treatment w/Doppler
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20032561
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cerebral Artery Syndrome; Anterior Cerebral Artery Stroke; Acute Ischemic Stroke; Coronary Artery Disease; Cardioembolic Stroke; Congestive Heart Failure; Diabetes; Vasogenic Cerebral Edema
Keywords: systolic blood pressure; Transcranial Doppler
MeSH Terms: conditions — Infarction, Anterior Cerebral Artery; Ischemic Stroke; Coronary Artery Disease; Embolic Stroke; Heart Failure; Diabetes Mellitus; Brain Edema

STUDY DESIGN:
Intervention Model Description: Prospective single center observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anterior circulation stroke that underwent EVT including tandem occlusions (Experimental): Subjects with anterior circulation stroke including ACA, MCA or ICA stroke that underwent EVT including tandem occlusions
  Interventions: Other: TCD measurement; Other: TCD parameters; Other: Baseline characteristics; Other: Clinical data will be collected; Other: All follow-up patients receive a phone call

INTERVENTIONS:
Other: TCD measurement — TCD measurement will be collected with TCD low frequency MHz probes. All TCD operations will be performed by a trained sonographer to assess bilateral MCA, ACA, PCA, Siph, and OA. TCD examinations will be performed as soon as possible after EVT, daily for 3 days and, when possible, as close to any reported neurological deterioration or CT brain scan performed within 72 hours of EVT.
Other: TCD parameters — TCD parameters are PSV, EDV, MFV, and PI. Sampling volume will be 5-10 mm, and the monitoring depth on transtemporal windows will be adjusted to gather appropriate vessel segment, e.g. 20-30 mm in the leptomeningeal flow, 40-50 mm in the distal MCA, 50-60 mm in the proximal MCA, 70-75 mm in the ACA, 62-70 mm in PCA, and transorbital, including 60-64 mm in the Siph and 50-60 mm in the OA. TAMMV and PI will be automatically derived from preset.
  Additionally, flow diversion will be assessed as an indirect indicator of arterial occlusion or severe stenosis in the middle cerebral artery (M1). It will be identified by TCD based on the following criteria: (1) low-resistance flow pattern in the anterior or posterior cerebral artery, and (2) mean flow velocity in the ACA or PCA greater than or equal to that in the MCA.
Other: Baseline characteristics — Baseline characteristics will be collected, including age, sex, ethnicity, history of HTN, DM, DLP, CHF, AF, CA, CKD, previous CAD, cirrhosis, mRS, previous stroke or TIA, current antiplatelet usage, current anticoagulant usage, smoking, and alcohol status. This data will be collected through a combination of verbal interviews with participants/LAR legally authorized representatives and a review of their medical history charts.
Other: Clinical data will be collected — Clinical data will be collected, including blood pressure values before, during, and after TCD as well as, Door to needle, Door to groin, Groin to first pass, time from recanalization to TCD, baseline NIHSS, site of occlusion, infarct core volume, mismatch volume, mismatch ratio, and IVT treatment status. Classification of stroke etiologies will be collected based on widely accepted TOAST criteria categorized in large vessel atherosclerosis (LAA), cardio-embolism (CE), small vessel occlusion (SAO), Stroke of other determined etiology (SOC), and stroke of undetermined etiology (SUC) [30]. This data will be collected by reviewing medical charts from EHR coded as part of standard care.
Other: All follow-up patients receive a phone call — All follow-up patients receive a phone call as part of standard post thrombectomy care from the stroke nurses to gather modified Rankin Scale at 7 days and 90 days since hospital discharge.

SUMMARY:
Endovascular therapy (EVT) has proven to be more beneficial for patients with AIS caused by large vessel occlusions (LVO) than medical management alone. A recent meta-analysis of 5 RCTs showed that EVT significantly reduced disability at 90 days compared to medical management [1]. Despite its obvious benefits, patients may have neurological deterioration despite successful thrombectomy due to ischemia progression, intracranial hemorrhage, re-occlusion, or vasogenic edema. The incidence of early neurological deterioration (END) following EVT for acute stroke has been reported to be ranging from 14.1-35.2% with some studies defining END up to 7 days and some restricting the definition between 6-72 hours post thrombectomy. A small proportion of these patients, approximately 5.9-10.5%, experienced sICH following EVT. Whether END occurs due to ischemic or hemorrhagic it leads to worse outcomes.

DETAILED DESCRIPTION:
One reason for END is impaired cerebral autoregulation (CAR), subsequent to the LVO. Cerebral autoregulation (CAR) is the brain's ability to maintain relatively constant cerebral blood flow (CBF) despite fluctuations in systemic blood pressure. Failure of CAR is associated with secondary brain injury that may occur as an extension of the initial ischemic core with the no-reflow phenomenon in hypoperfusion. CAR may also be impaired causing cerebral edema, or hemorrhagic transformation with cerebral hyperperfusion. The degree of recanalization, preexisting hypertensive profile and post thrombectomy blood pressure can impact CAR and contribute to risk of hypo or hyperperfusion. In the DAWN trial, EVT was performed 6 to 24 hours after stroke onset, and BP was controlled to less than 140/90 mmHg in patients who achieved reperfusion with mTICI 2b or 3. This trial reported incidents of 6% for END and 14% for sICH, respectively. The BEST-II trial, which compared moderate BP control (SBP of either 140 or 160 mmHg) with standard control (SBP less than 180 mmHg) in patients successful post-EVT, suggested a low probability of benefit from lower SBP targets. The incidence of sICH in this trial was 5%. The 2019 American Heart Association/American Stroke Association (AHA/ASA) guidelines recommended a BP goal of 180/105 after EVT, as a reasonable extrapolation from the IVT literature. However, the recommendation for BP control still lacks clear supporting evidence. While the proposed role of CAR in post thrombectomy underscores the need for evaluating CAR in patients after EVT to evaluate patient specific systemic blood pressure parameters bedside measurements of CAR in these patients is still not a practical clinical possibility. Most CAR evaluation devices need ICP that is invasive and typically not amenable in post thrombectomy patients. Non-invasive methods of evaluating CAR based on transfer function analysis are still not validated for widespread clinical use and need significant IT infrastructure.

TCD is recognized as a diagnostic tool for measuring CBF. One of its key advantages lies in its ability to perform non-invasive, real-time monitoring directly at the patient's bedside, making it invaluable in acute stroke management. TCD based CBV measurement can provide valuable insights into cerebral hemodynamics and when combined with systemic BP data TCD has the potential to guide critical decisions, such as post-EVT BP management, to prevent secondary injuries like ICH. Tools like TCD, which can provide real-time assessment of cerebral hemodynamics, remain underutilized in this context. We propose this study to evaluate specific TCD parameters in post-EVT patients who develop early neurological deterioration or ICH that can serve as future targets of therapy. Understanding these parameters may provide valuable insights into the hemodynamic changes that occur after EVT and help guide future BP management strategies to reduce the risk of complications like ICH.

ELIGIBILITY:
Inclusion Criteria:

* Anterior circulation stroke including ACA, MCA or ICA stroke that underwent EVT including tandem occlusions.
* Age ≥ 18 years

Exclusion Criteria:

* Difficulty in detecting the acoustic window by TCD
* Pregnancy
* Incarcerated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2027-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Determine correlation between transcranial Doppler (TCD) parameters | Within 72 hours of any large vessel occlusion
  Compare peak flow velocity, mean flow velocity, and pulsatility index. Transcranial Doppler (TCD) ultrasound uses sound waves to measure blood flow in the brain's arteries, providing scores that indicate normal flow or potential issues like vasospasm or increased stroke risk. Normal TCD scores for the middle cerebral artery (MCA) range from 55 cm/sec for normal flow, with elevated velocities indicating mild to severe vasospasm.

SECONDARY OUTCOMES:
Discharge Disposition | Study Duration, 24 months
  Discharge disposition (discharge to home, acute rehabilitation, skilled nursing facility, long-term acute care facility, hospice/palliative care/death). It is the final place or setting to which the patient was discharged on the day of discharge.
Modified Rankin Scale | 3 months
  Modified Rankin scale closest to 3 months. The Modified Rankin Scale (mRS) is a 6-point disability scale used to measure the degree of disability or dependence in activities of daily living after a stroke or other neurological disability. It is a widely used outcome measure in stroke clinical trials and clinical care. 0-2: Indicate mild to moderate disability, with patients being largely independent. 3-5: Indicate moderate to severe disability, requiring assistance with daily activities. 6: Indicates death.
Interaction between collateral circulation status and mean arterial pressure | 72 hours
  To investigate the interaction between collateral circulation status and mean arterial pressure (MAP) in relation to predicting risk of END within 72 hours. In the context of cerebral stroke, the relationship between collateral circulation status and mean arterial pressure (MAP) is complex and significant. Poor collateral circulation, particularly in the case of acute large vessel occlusion (LVO), increases the dependence of blood flow on MAP. Cerebral autoregulation, the brain's ability to maintain constant blood flow despite changes in MAP, is impaired during LVO. This means that even within the typical autoregulation range (50-150 mmHg), the brain's ability to compensate for blood pressure fluctuations is reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sarwal, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States